CLINICAL TRIAL: NCT02487758
Title: Ridge Preservation Comparing the Clinical and Histologic Healing of Flap vs. Flapless Approach to Grafting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Graduate Periodontics Director, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15.0531
Record Dates: First submitted 2015-06-19; First posted 2015-07-01 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ridge preservation Flap (Experimental): The flap procedure will consist of a full-thickness papilla preservation flap performed on the buccal and a full thickness flap on the palatal.
  Interventions: Procedure: Ridge Preservation
- Ridge preservation Flapless (Experimental): The test will be a flapless technique with tunneling and an intramucosal vertical incision on the buccal.
  Interventions: Procedure: Ridge Preservation

INTERVENTIONS:
Procedure: Ridge Preservation — Ridge Preservation Comparing the Clinical and Histologic Healing of Flap vs. Flapless Approach to Grafting

SUMMARY:
Ridge Preservation Comparing the Clinical and Histologic Healing of Flap vs. Flapless Approach to Grafting

DETAILED DESCRIPTION:
Thirty patients will be treated using the principles of guided bone regeneration and ridge preservation. Fifteen test patients will receive the flapless technique with an intrasocket cancellous cortical particulate allograft plus a facial overlay graft using a bovine xenograft plus Alloderm GBR. The positive control group of fifteen patients will receive the flap technique with an intrasocket cancellous cortical particulate allograft plus a facial overlay graft using a bovine xenograft plus Alloderm GBR. Approximately, four months post-surgery, a trephine core will be taken from the grafted site immediately prior to implant placement and submitted for histologic processing.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy male or female who is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Presence or history of osteonecrosis of jaws.
3. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of duration.
4. Patients who have been treated with oral bisphosphonates for more than three years.
5. Patients with an allergy to any material or medication used in the study.
6. Previous head and neck radiation therapy.
7. Chemotherapy in the previous 12 months.
8. Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change in post-extraction site to 4 month change in crestal osseous width | 4 months
  Changes in post-extraction to 4 month change in ridge measurements at the mid-defect alveolar crest and 5 mm apical taken with a caliper.

SECONDARY OUTCOMES:
Change in Soft tissue thickness | 4 months
  Soft tissue thickness measurements taken with a #40 endodontic reamer.
Percent osseous tissue | 4 months
  A trephine core will be harvested at 4 months. Following histologic processing the osseous core will be classified into percent vital bone, nonvital bone and trabecular space.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville